CLINICAL TRIAL: NCT07005635
Title: Comparison of The Effects of Different Time Reminder on Surgical Hand Scrub: A Randomized Controlled Study
Brief Title: The Effects of Different Time Reminder On Surgical Hand Scrubing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Ozgu Bakcek, Associate professor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: YuksekIhtisass
Record Dates: First submitted 2025-05-12; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Surgical Site Infection
Keywords: Surgical Hand scrub; skill laboratory; satisfaction; Time reminder
MeSH Terms: conditions — Surgical Wound Infection; Personal Satisfaction | interventions — Clinical Alarms

STUDY DESIGN:
Intervention Model Description: Music group Alarm group Control group
Who Masked: Participant
Masking Description: While operating room services program students scrubing hands in School skill laboratory during hand scrubing music group, listen to music at the end of the scrubing alarm group, listen alarm sound and the control group follows scrubing time on a washing cabin clock
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music group (Experimental): While operating room services program students scrubing hands in School skill laboratory during hand scrubing music group, listen to music
  Interventions: Other: Listening Music
- Alarm group (Experimental): While operating room services program students scrubing hands in School skill laboratory at the end of the scrubing alarm group, listen alarm sound
  Interventions: Other: Alarm
- Control group (No Intervention): While operating room services program students scrubing hands in School skill laboratory the control group follows scrubing time on a washing cabin clock

INTERVENTIONS:
Other: Listening Music — Music group students listen Beethoven Moonlight Sonata during scrubing hands
  Other Names: Beethoven Moonlight Sonata
  Arms: Music group
Other: Alarm — Alarm group students listen alarm sound at the end of the (2 min) during scrubing hands
  Other Names: Alarm sound
  Arms: Alarm group

SUMMARY:
When surgical hand scrubing is not done properly, it can negatively affect patient outcomes. In addition to the entire surgical team being able to perform surgical hand scrubing properly, every student studying in the health field who will work in operating rooms should also learn and practice surgical hand washing correctly. In this context, this study aims to evaluate the satisfaction and success of different time reminder systems on students' surgical hand scrubing skills.

DETAILED DESCRIPTION:
This randomized controlled study will carry out Sixty-six (music group= 22, alarm group= 22, control group= 22) first year undergraduate operating room services program students. This program places at a Vocational School of Health Services, Operating Room Services Programme in Ankara Turkey.

ELIGIBILITY:
Inclusion Criteria:

* to be a first-year students of the operating room services program
* to be volunteered

Exclusion Criteria:

* previous experience working in the operating room

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Surgical Hand Scrub Time | 3 months
  Second during surgical hand scrubbing

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Özgü Bakçek, Ankara, Eyalet/Yerleşke
  - Yuksek Ihtisas University, Ankara

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Spruse, L. (2013). Back to basics: Hand hygiene and isolation. AORN Journal, 98(5), 449-460. — http://doi.org/10.1097/QCO.0000000000000080
- See also: NICE. (2020). Surgical site infections: prevention and treatment CG74. Clinical Guideline-National Insitute of Health and Care Excellence, April 2019, 1-29. — http://www.nice.org.uk/guidance/ng125
- See also: Msosa, A., Bruce, J., & Crouch, R. (2021). Effect of a formative assessment intervention on nursing skills laboratory learning in a resource-constrained country. Nurse Education Today, 97, 104677. — http://doi.org/10.1016/j.nedt.2020.104677
- See also: Kilic, S. (2015). Kappa test. Journal of Mood Disorders, 5(3), 142. — http://doi.org/10.5455/jmood.20150920115439
- See also: Ince, S., & Çevik, K. (2017). The effect of music listening on the anxiety of nursing students during their first blood draw experience. Nurse Education Today, 52, 10-14. — http://doi.org/10.1016/j.nedt.2017.02.009
- See also: Faul, F., Erdfelder, E., Lang, A. G., & Buchner, A. (2007). G*Power 3: A flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behavior Research Methods, 39(2), 175-191. — http://doi.org/10.3758/BF03193146
- See also: CDC. (2002). Guidelines for hand hygiene in healthcare settings. CDC Morbidity and Mortality Weekly Report, 51(RR-16). — http://doi.org/10.1097/01.idc.0000129851.34508.48
- See also: Bakcek, O., Tastan, S., Iyigun, E., Kurtoglu, P., & Tastan, B. (2020). Comparison of PechaKucha and traditional PowerPoint presentations in nursing education: A randomized controlled study. Nurse Education in Practice, 42(January), — http://doi.org/10.1016/j.nepr.2020.102695
- See also: akcek Akcelik, O. B., Ayhan, H., & Tastan, S. (2023). Comparison of the Effects of Body Mechanics Education Methods on Pain, Disability, and Quality of Life: A Randomized Controlled Study. Pain Management Nursing, 24(6), e152-e159. — http://doi.org/10.1016/j.pmn.2023.08.009
- See also: Baghbaninaghadehi, F., Armijo-Olivo, S., & Woodhouse, L. (2016). Fundamentals of Randomization in Clinical Trial. International Journal of Advanced Nutritional and Health Science, 4(1), 174-187. — http://doi.org/10.23953/cloud.ijanhs.143